CLINICAL TRIAL: NCT00524784
Title: Phase 1/2a, Multicenter, Open-Label Study Designed to Evaluate the Safety, Tolerability and Preliminary Efficacy of ApoCell Administration, a Donor Apoptotic Cell-Based Product, for the Prevention of Acute Graft Versus Host Disease (GvHD) in Subjects With Hematologic Malignancies Undergoing Allogeneic Sibling HLA-Matched Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Open-Label Study Designed to Evaluate the Safety and Preliminary Efficacy of ApoCell for the Prevention of Acute GvHD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TLX-APO-101IL-HMO-CTIL
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Graft Versus Host Disease; Hematological Malignancies
Keywords: GVHD; HSCT; BMT; APOPTOTIC CELLS
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Three subjects per cohort will be treated with ApoCell according to an escalating schedule of doses
  Interventions: Biological: ApoCell

INTERVENTIONS:
Biological: ApoCell — Three subjects per cohort will be treated with ApoCell according to an escalating schedule of doses starting at a single dose of 35 million apoptotic cells/kg in the first cohort of three subjects. Unless a DLT is experienced by subjects in a given cohort, the dose in the subsequent cohort will be increased by two-fold. The second cohort will receive 70 millions cells/kg, and the third cohort 140 millions cells/kg. The final fourth cohort will receive 210 millions cells/kg.

SUMMARY:
Bone marrow transplantation (BMT) has revolutionized the treatment of hematopoietic malignancies.Unfortunately, graft versus host disease (GvHD) remains a major toxicity that greatly limits the application and efficacy of BMT.Current standard prophylaxis and therapy for acute GvHD include mainly the use of immunosuppressive drugs that help less than 50% of the patients and are associated with increased infection risk. ApoCell treatment is anticipated to be a prophylactic measure for acute GvHD by inducing tolerance in the donor effector cells, leading to a potentially significant decrease in GVHD.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem-cell transplantation (HSCT) has revolutionized the treatment of hematopoietic malignancies, inherited hematopoietic disorders, aplastic anemia, and other severe diseases. Unfortunately, graft versus host disease (GvHD) remains a major toxicity that greatly limits the application and efficacy of allogeneic HSCT, occurring commonly after the procedure and affecting 30 to 80% of patients. Acute GvHD occurs within 100 days in up to 50% of allogeneic HLA-matched HSCT recipients despite prophylactic immunosuppressive drugs.

The most efficient treatment for GvHD prevention is T cell depletion. However, most clinicians avoid that modality due to the crucial effect of T cells in prevention of tumor relapse. Current standard prophylaxis and therapy for acute GvHD include mainly the use of immunosuppressive drugs that help less than 50% of the patients and are associated with increased infection risk. New strategies of GvHD prophylaxis are examined and this study uses a physiological strategy of antigen presenting cell (APC) tolerance induction that will modulate effector cells either directly or via T regulatory cells.

ApoCell treatment is anticipated to be a prophylactic measure for acute GvHD by inducing tolerance in the donor effector cells, leading to a potentially significant decrease in the immune response of the donor cells against the recipient. The effects of apoptotic cells on preventing GvHD may involve the following mechanisms: inhibit pro-inflammatory cytokine production, promote anti-inflammatory cytokines production, induce tolarogenic APCs, decrease ability to stimulate T-cell responses, delete CD8 T-effector cells, induce regulatory T-cells, and inhibit response to inflammatory cytokines and LPS.

Tolarex Ltd. is proposing a novel cell-based approach of donor apoptotic cells treatment, ApoCell, for a Phase I-IIa study of patients undergoing sibling HSCT with high risk of developing acute GvHD. The ApoCell product is composed of HLA-matched donor mononuclear enriched leukocytes in the form of liquid suspension that will be injected intravenously to the patient 24 hours prior to HSCT. The ApoCell suspension contains at least 55% of early apoptotic cells. The cell suspension is prepared under cGMP conditions with PBS solution within 8 hours prior to intravenous injection and should be stored at 2-8oC until administered.

ELIGIBILITY:
Inclusion Criteria: Recipient

1. Adult male or female subjects, 18-60 years of age, inclusive, at the time of screening visit weighing at least 40 kg.
2. Subjects are eligible for allogeneic sibling HLA-matched HSCT for any disease for which transplantation is appropriate except progressive or poorly controlled malignancies. Only one of the following malignancies should be present:

   1. Acute lymphoblastic leukemia or acute myeloid or undifferentiated or biphenotypic, leukemia, in complete remission or beyond but with ≤10% blasts in bone marrow.
   2. Acute myeloid leukemia in complete remission if it has evolved from myelodysplastic syndrome (MDS) (there should be documented diagnosis of MDS at least 3 months prior to diagnosis of acute myeloid leukemia).
   3. Myelodysplastic syndromes - MDS
   4. Therapy related MDS (irrespective of IPSS).
   5. Chronic myeloid leukemia (CML) chronic phase-1 (imatinib failures, imatinib intolerance), or any CML beyond first chronic phase.
   6. Multiple Myeloma.
3. The donor and recipient must have at least a 7/8 HLA match at the HLA A, B, C, and DR loci.
4. Life expectancy of at least 6 months at the time of the baseline visit.
5. Karnofsky performance status score ≥ 80% at time of the screening visit.
6. Cardiac left ventricular ejection fraction ≥ 40% in adults within 4 weeks of initiation of conditioning; required if prior anthracycline exposure or history of cardiac disease.
7. Pulmonary function test with DLCO, FEV1 and FVC of ≥ 60%.
8. Oxygen saturation ≥ 90% on room air.
9. Subjects must have normal organ function as defined below:

   1. AST (SGOT)/ALT (SGPT) ≤ 2.5 x upper limit of normal (ULN).
   2. Serum creatinine <2.5 mg/dL.
   3. Serum bilirubin <3 mg/dL.
   4. Coagulation markers - PT and PTT within normal limits.
10. Signed written informed consent to participate in the study independently by subject. Subjects requiring a guardian to sign informed consent will not be included.
11. Ability to comply with the requirements of the study.
12. If female, agree to use an acceptable method of birth control or be surgically sterile, and have a negative pregnancy test regardless of child-bearing potential.

Exclusion Criteria: recipient

1. Participation in an investigational trial within 30 days of the screening visit.
2. Have progressive or poorly controlled malignancies.
3. T-cell depleted allograft.
4. Uncontrolled infections including sepsis, pneumonia with hypoxemia, persistent bacteremia, or meningitis within two weeks of the screening visit.
5. Current known acute or chronic infection with HBV or HCV.
6. Known human immunodeficiency virus (HIV) infection or AIDS.
7. Subjects with severe or symptomatic restrictive or obstructive lung disease or respiratory failure requiring ventilator support.
8. Subjects with other concurrent severe and/or uncontrolled medical condition which could compromise participation in the study (i.e. active infection, uncontrolled diabetes, uncontrolled hypertension, congestive cardiac failure, unstable angina, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within six months, chronic liver or renal disease, active upper gastrointestinal tract ulceration).
9. Any chronic or acute condition susceptible of interfering with the evaluation of investigational product effect.
10. Any form of substance abuse (including drug or alcohol abuse), psychiatric disorder or any chronic condition susceptible, in the opinion of the investigator, of interfering with the conduct of the study.
11. Organ allograft or previous history of allogeneic stem cell transplantation.
12. For all women: A positive pregnancy test at screening or breast-feeding.
13. Subjects who are likely to be non-compliant or uncooperative during the study.

Inclusion criteria: Donor

1. Male or female donors, 18 - 65 years of age, inclusive.
2. The donor and recipient must have at least a 7/8 HLA match at the HLA A, B, C, and DR loci.
3. Above 40 kg.
4. Not pregnant and negative pregnancy test.
5. Serum creatinine < 2.5 mg/dL.
6. Oxygen saturation ≥ 90% on room air.
7. No severe or symptomatic restrictive or obstructive lung disease or respiratory failure requiring ventilator support.
8. No uncontrolled hypertension or congestive heart failure, active angina pectoris requiring the use of nitrates, or major ventricular arrhythmia or cardiac failure requiring active treatment.
9. Not HIV-1/2 or HTLV I/II seropositive or evidence of acute CMV infection.
10. Not seropositive for Hepatitis B or C.
11. Not positive for syphilis.
12. No known bone marrow disease.
13. No significant organ dysfunction.
14. No acute infectious disease within two weeks of donation.
15. Willingness to donate hematopoietic blood mononuclear cells for the generation of ApoCell more than one time if required and in addition to the donation for the HSCT.
16. Ability to provide written informed consent and comply with study requirements.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-12 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Determine the safety profile and tolerability [dose limiting toxicity (DLT)] of ascending doses of ApoCell in subjects undergoing allogeneic sibling HLA-matched HSCT within 180 days post-transplantation. | 180 days

SECONDARY OUTCOMES:
*Determine the success rate for HSC engraftment and time to successful engraftment. *Describe the rates and grade of acute GvHD following ApoCell infusion. *Determine the success rate for HSC engraftment and time to successful engraftment. *Determine | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Reuven Or, Professor, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Department of Bone Marrow Transplantation, Jerusalem, Israel

REFERENCES:
- [Derived] Mevorach D, Zuckerman T, Reiner I, Shimoni A, Samuel S, Nagler A, Rowe JM, Or R. Single infusion of donor mononuclear early apoptotic cells as prophylaxis for graft-versus-host disease in myeloablative HLA-matched allogeneic bone marrow transplantation: a phase I/IIa clinical trial. Biol Blood Marrow Transplant. 2014 Jan;20(1):58-65. doi: 10.1016/j.bbmt.2013.10.010. Epub 2013 Oct 15. PMID 24140121